CLINICAL TRIAL: NCT01607528
Title: Probiotic Modulation of Gut Microflora in Cirrhosis: Influence on Immune Function and Infections
Brief Title: Influence of Probiotics on Infections in Cirrhosis
Acronym: PIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PIC-2010
Record Dates: First submitted 2012-04-13; First posted 2012-05-30 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Active Comparator): 6 g of Winclove-849 containing Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus salivarius W24, Lactococcus lactis W19, Lactococcus lactis W58 at a concentration of 2.5 x 10E9 cfu/g per day
  Interventions: Dietary Supplement: Winclove-849
- Placebo (Placebo Comparator): A similar looking and tasting powder
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Winclove-849 — 6 g of Winclove-849 containing Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus salivarius W24, Lactococcus lactis W19, Lactococcus lactis W58 at a concentration of 2.5 x 109 cfu/g
  Arms: Probiotic
Dietary Supplement: Placebo — A similar looking and tasting powder with no active substances
  Arms: Placebo

SUMMARY:
Liver cirrhosis is the 10th most common cause of death in the western world. Infection is the most common precipitant of deterioration of liver function in cirrhosis. Endotoxin, derived from gram-negative organisms in the gut, can enter the circulation due to increased gut permeability and contributes to neutrophil dysfunction, infection risk and mortality in alcoholic cirrhotics. As probiotics decrease gram-negative organisms in the gut and/or decrease gut permeability, the investigators hypothesize that probiotic treatment would restore neutrophil function and prevent infection in alcoholic cirrhosis.

The investigators hypothesize that administration of a probiotic mixture in patients with liver cirrhosis will improve innate immune function through alteration of the gut bacterial flora and gut barrier integrity.

The aim of this randomised, double-blinded placebo-controlled study is to assess whether food supplementation with probiotic mixture improves neutrophil phagocytic capacity in patients with cirrhosis and decreases the incidence of significant infections.

92 patients with alcoholic cirrhosis will be included according to a sample size calculation from preliminary data. Patients will be randomized in two groups: Group 1 receives a probiotic mixture Group 2 receives a similar looking and tasting placebo without bacteria. The recruited patients will be treated for 6 months. Besides routine clinical and laboratory assessments, neutrophil function, toll-like receptor expression, endotoxin levels, bacterial DNA, cytokine levels, albumin oxidation, gut permeability and analysis of gut microflora will be performed. Furthermore nutritional status and quality of life will be assessed.

Primary endpoints will be neutrophil phagocytosis. Secondary endpoints will be significant infection, neutrophil oxidative burst, neutrophil toll-like receptor expression, endotoxin levels, bacterial DNA; cytokine levels, albumin oxidation, gut barrier function and bacterial flora, nutritional status and quality of life.

If our hypothesis holds true, probiotics will provide an easily applicable and cost effective method to improve immune function and to prevent infection in liver cirrhosis. It is possible that this can improve survival of patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria: • Patients aged between 18-80 years

* Clinical and radiological evidence of cirrhosis, and/or biopsy proven liver cirrhosis of any cause
* Informed consent

Exclusion Criteria:

* Child-Pugh score > 11
* Abstinence from alcohol for < 2 weeks at the time of screening for inclusion
* Clinical evidence of active infection
* Antibiotic treatment within 7 days prior to enrolment
* Gastrointestinal haemorrhage within previous 2 weeks
* Use of immunomodulating agents within previous month (steroids etc.)
* Use of proton pump inhibitors for preceding two weeks
* Concomitant use of supplements (pre-, pro-, or synbiotics) likely to influence the study
* Renal failure (such as hepatorenal syndrome), creatinine >1.7 mg/dL
* Hepatic encephalopathy II to IV
* Pancreatitis
* Other organ failure
* Hepatic or extra-hepatic malignancy
* Pregnancy
* Presumed non-compliance to the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in neutrophil phagocytic capacity | Change from baseline to 6 months
  Percentage of neutrophil granulocytes showing phagocytosis of FITC (fluorescein isothiocyanate) -labelled E.coli bacteria

SECONDARY OUTCOMES:
Number of clinically significant infections | during 12 months
  Occurence of infections that require specific treatment and/or hospitalisation during the study period of 12 months
endotoxin levels | 0, 6, 12 months
  Endotoxin in serum (EU/ml)
neutrophil oxidative burst | 0, 6, 12 months
  percentage of neutrophil granulocytes showing oxidative burst with and without stimulation and mean fluorescence activity
neutrophil toll like receptor expression | 0, 6, 12 months
  percentage of neutrophil granulocytes showing TLR (Toll-like receptor) 2, TLR4 or TLR9 expression and mean fluorescence activity
albumin oxidation | 0, 6, 12 months
  oxidative status of albumin in the plasma (percentage of (human mercaptalbumin) HMA, (human non-mercaptalbumin) HNA1 and HNA2)
inflammatory response | 0, 6, 12 months
  elevation of one or more inflammatory markers: C reactive protein (mg/ml), lipopolysaccharide binding protein (ng/ml), soluble CD (cluster of differentiation) 14 (ng/ml)
bacterial flora | 0, 6, 12 months
  isolation of bacterial DNA and sequencing the gut microbiome from stool and duodenal aspirate
quality of life | 0, 6, 12 months
  (short form) SF-36 questionaire
nutritional status | 0,6, 12 months
  subjective global assessment
changes in gut permeability over time | 0, 6, 12 months
  elevated lactulose mannitol ratio, elevated zonulin

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer-Köllner, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Geraz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Egger M, Horvath A, Pruller F, Fickert P, Finkelman M, Kriegl L, Gronbaek H, Moller HJ, Prattes J, Krause R, Hoenigl M, Stadlbauer V. Fungal translocation measured by serum 1,3-ss-D-glucan correlates with severity and outcome of liver cirrhosis-A pilot study. Liver Int. 2023 Sep;43(9):1975-1983. doi: 10.1111/liv.15648. Epub 2023 Jun 19. PMID 37334864
- [Derived] Stadlbauer V, Komarova I, Klymiuk I, Durdevic M, Reisinger A, Blesl A, Rainer F, Horvath A. Disease severity and proton pump inhibitor use impact strongest on faecal microbiome composition in liver cirrhosis. Liver Int. 2020 Apr;40(4):866-877. doi: 10.1111/liv.14382. Epub 2020 Jan 24. PMID 31943691